CLINICAL TRIAL: NCT01743924
Title: Bioavailability of Bioactive Compounds in Broccoli
Brief Title: Bioavailability of Chemopreventive and Nutritional Compounds in Broccoli
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universidad Politécnica de Cartagena (Other)
Collaborators: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Principal Investigator, Ginés Benito Martínez Hernández, Doctor, Universidad Politécnica de Cartagena
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: Broccoli_Bioav.
Record Dates: First submitted 2012-11-30; First posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Bioavailability
Keywords: Broccoli; Isothiocyanates; Pharmacokinetics; Sulforaphane; Myrosinase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raw (Experimental): Broccoli,200 grams
  Interventions: Other: raw broccoli
- cooked (Experimental): Microwaved, 200 grams
  Interventions: Other: raw broccoli

INTERVENTIONS:
Other: raw broccoli — To eat this plant material
  Other Names: Bimi; Kailan hybrid

SUMMARY:
The aim of this study was to determine the absorption of isothiocyanates (ITC) after ingestion of kailan-hybrid broccoli through the analysis of the correspondent urinary biomarkers. Furthermore, the effect of cooking (microwave) on the mentioned metabolic fate of these ITC was studied comparing to the uncooked vegetable.

DETAILED DESCRIPTION:
Background Glucosinolates (sulphur-containing compounds) are hydrolyzed by the plant enzyme myrosinase to ITC, which have chemopreventive properties. No information has been reported about the metabolic fate of ITC in the kailan-hybrid broccoli, which physicochemical characteristics could greatly influence that metabolic fate. Previous studies have shown that cooking process of vegetables may vary the human absorption of the correspondent nutritional and bioactive compounds.

Research Methods & Procedures A cross-over-design study of 7 subjects after ingestion of 200-g raw or microwaved kailan-hybrid broccoli was conducted. Total ITC equivalents in the vegetable, urine and blood samples were determined by HPLC as the cyclocondensation product of 1,2-benzenedithiol.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a body mass index between 19 and 28.
* Subjects age: 22-50 years-old.
* Good health of subjects: confirmed by medical history, physical examination and clinical laboratory analysis of urine and blood (complete blood count and liver function markers including serum glutamic-pyruvic transaminase bilirubin test and glucose-6-phosphate dehydrogenase).

Exclusion Criteria:

* Tobacco smoking.
* Use of regular medications.
* Had taken antibiotics for 4 weeks immediately preceding the study.
* History of kidney stones, diabetes mellitus, bleeding disorders or family history of iron overload/hemochromatosis.

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2011-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Metabolic fate of ITC of the kailan-hybrid broccoli after human comsuption | Up to 4 weeks
  Glucosinolates (sulphur-containing compounds) are hydrolyzed by the plant enzyme myrosinase to isothiocyanates (ITC), which have chemopreventive properties. Previous studies have shown that cooking process of vegetables may vary the human absorption of the correspondent nutritional and bioactive compounds.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Concepcion Maeztu Sardiña, Doctor, Study Chair — Comité ético de investigación clínica
Locations (1):
- Hospital General Universitario Reina Sofía, Murcia, Murcia, Spain